CLINICAL TRIAL: NCT04214236
Title: Evaluation of ciNPT Effects on Healing and Post-surgical Complications in High-risk Post- Bariatric Patients Undergoing Body-contouring Abdominoplasty: a Monocentric Prospective RCT
Brief Title: CiNPT for Abdominoplasties in Post-bariatric Patients Study
Acronym: CAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera, Ospedale Civile di Legnano (Other)
Collaborators: Acelity (Other)
Responsible Party: Principal Investigator, Silvio Abatangelo, Plastic Surgeon - Physician, Azienda Ospedaliera, Ospedale Civile di Legnano
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAPS/01
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Obesity, Morbid; Obesity; Obesity, Abdominal; Wound; Wound Infection; Wound Complication; Wound Dehiscence; Wound Contamination; Wound Heal; Wound; Abdomen; Incision; Incision Site Rash; Incision Site Bleeding; Incision Site Swelling; Incision Site Haematoma; Incision Site Infection; Incision Site Inflammation; Incision Site Complication; Incision Surgical; Surgery--Complications; Surgical Wound Infection; Surgical Site Infection; Scarring as Surgical Complication; Scar; Scarring
Keywords: Closed-incision negative pressure therapy; Negative pressure wound therapy; Wound care; Surgical incision; Wound complication; Dehiscence; Surgical Site Infection; Seroma; Hematoma; Wound Healing; Inflammation; Incisional Wound; Abdominoplasty; Abdominal panniculectomy; Body contouring
MeSH Terms: conditions — Obesity, Morbid; Obesity; Obesity, Abdominal; Wounds and Injuries; Wound Infection; Abdominal Injuries; Surgical Wound; Surgical Wound Infection; Cicatrix; Seroma; Hematoma; Inflammation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Case-control Experimental/Interventional Group: post-operative ciNPT (first 7 days) Control Group: post-operative standard wound care
Who Masked: Outcomes Assessor
Masking Description: Analysis of data and statistical analysis will be blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ciNPT group (Experimental): Subjects will receive post-operative incisional wound care by ciNPT (125 mmHg, continuous suction) for the first 7 days after surgery.
  Interventions: Device: ciNPT group
- Control group (Sham Comparator): Subjects will receive post-operative incisional wound care by standard non-adherent surgical dressing (vaseline petrolatum gauze),
  Interventions: Other: Control group

INTERVENTIONS:
Device: ciNPT group — Closed-incision negative pressure therapy (ciNPT) will be applied for 7 day using continuous suction at 125 mmHg. To deliver ciNPT we will use a commercially available, FDA-approved device, used according to the manufacturer' indications (PREVENA™ Incision Management System (KCI, San Antonio, Texas, USA). After the first 7 post-operative days, subjects will discontinue the ciNPT and follow a standard wound care protocol.
  Other Names: ciNPT; PREVENA™ Incision Management System; closed-incision negative pressure therapy
  Arms: ciNPT group
Other: Control group — Standard non-adherent surgical dressing (Vaseline petrolatum gauze) will be used for management of incisional wounds in the control group. Dressing changes will be performed per standard wound care protocol.
  Other Names: Standard incisional wound care
  Arms: Control group

SUMMARY:
The overarching goal of this research is to assess whether the post-operative use of closed-incision Negative Pressure Therapy (ciNPT) accelerates healing of surgical wounds, improves surgical outcomes, and reduces the rate of local complications in high-risk, obese, post-bariatric patients undergoing abdominal body-contouring procedures (abdominal panniculectomy or "abdominoplasty") compared to standard wound care.

The investigators postulate that ciNPT can cost-effectively improve outcomes and standard of post-surgical care in this specific category of patients.

This hypothesis will be tested through a prospective, interventional, case-control, randomized clinical trial.

DETAILED DESCRIPTION:
In the United States (US) 37% of the adult population is obese and 5% is considered morbidly obese. Similar trends have been observed in Europe and more recently in Asia. A large number of obese patients seeks treatment through bariatric surgery or diet-lifestyle changes. The resulting massive loss of weight leaves patients with an excess cutaneous tissue, requiring body-contouring procedures.

In the US 85% of post-bariatric patients seek body-contouring surgeries. Due to systemic and local factors, these procedures show a rate of local complications as high as 68-80%, significantly prolonging hospitalization and increasing treatment-related costs.

Several clinical studies have shown that external suction (Closed Incision Negative-Pressure Therapy, ciNPT) can accelerate closure of surgical wounds in patients at high-risk for impaired/delayed healing and can significantly reduce the rate of local complications. The investigators believe that ciNPT might significantly decrease the rate of minor local complications in post-bariatric patients undergoing body-contouring procedures, and that this strategy could represent a cost-effective adjuvant treatment in body-contouring procedures.

The investigators' preliminary study experience on post-bariatric obese patients undergoing an abdominoplasty and post-operatively treated with ciNPT, showed that ciNPT promotes effective and prompt wound closure minimizing peri-operative/post-operative complications in these patients. The investigators also showed that ciPNT positively impacts the length of hospitalization and the rate of secondary surgeries in these patients.

Based on this successful preliminary experience, the invetsigators here propose to validate these findings in a prospective RCT.

ELIGIBILITY:
Inclusion Criteria:

* previous bariatric surgery for weight loss
* candidate for/undergoing an abdominal panniculectomy (abdominoplasty)
* Residual BMI >30 kg/m2 at the time of the operation
* Evidence of pannus (abdominal) ptosis (Pittsburgh Rating Scale >2)
* Lipodystrophy and inelasticity of the skin
* Presence at the time of surgery of at least one local risk factor (e.g. a history or the presence of local complications such as skin blistering, recurrent erythema, panniculitis, or chronic infection; history of abdominal hernia or need for abdominal hernia repair) OR one systemic risk factor (diabetes, smoking habit, serum proteins below 6g/dL).

Exclusion Criteria:

* Severe systemic co-morbidities (defined as ASA III or higher)
* Malignant tumors
* Conditions or medications affecting wound healing (e.g. steroidal drugs or keloids)
* Known allergies to components of the treatment
* Presence of severe local cutaneous complications (open wounds, extensive infections) at the time of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of post-surgical local complications | 30 days
  The change in post-surgical local complications (Skin blistering/necrosis, Surgical Site Infections, hematoma, seroma, need for re-operation) through 30 days after surgery.

SECONDARY OUTCOMES:
Time-to-heal | <60 days
  A change in time (days) to complete wound closure for treated groups vs. controls.
Scar quality: Vancouver Scar Scale | 30 and 90 days
  A change in the macroscopic quality of scars at a 30 and 90 days follow up (measured with the Vancouver Scar Scale-VSS [Score range: 0-13, lower scores being a better outcome]).
Medical costs | 60 days
  A change in direct medical costs (considering cumulative costs related to: hospitalization, standard and additional post-operative care, additional surgical and medical care for complications) in the first 60 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Abatangelo, M.D., Principal Investigator — ASST Ovest Milanese

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Result] Abatangelo S, Saporiti E, Giatsidis G. Closed Incision Negative-Pressure Therapy (ciNPT) Reduces Minor Local Complications in Post-bariatric Abdominoplasty Body Contouring: a Retrospective Case-Control Series. Obes Surg. 2018 Jul;28(7):2096-2104. doi: 10.1007/s11695-018-3279-8. PMID 29730777